CLINICAL TRIAL: NCT02523521
Title: Impacte d'un Programa d'Exercici Per Nens d'Entre 4 a 6 Anys Amb Displàsia Broncopulmonar
Brief Title: Impact of an Exercise Program for Children Aged 4 to 6 Years With Bronchopulmonary Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Nens de Barcelona (Other)
Responsible Party: Principal Investigator, Morales, physiotherapist, Hospital de Nens de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PIC-140-15
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Bronchopulmonary Dysplasia; Healthy
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bronchopylmonary Dysplasia Control (No Intervention): Nothing
- Bronchopylmonary Dysplasia Intervention (Experimental): physical activity program.
  Interventions: Behavioral: Physical activity program
- Healthy children (No Intervention): Nothing.

INTERVENTIONS:
Behavioral: Physical activity program — physical activity program for a bronchopulmonary dysplasia children.
  Arms: Bronchopylmonary Dysplasia Intervention

SUMMARY:
The purpose of this study is to determine the effects of a physical activity program for children with Bronchopulmonary Dysplasia.

DETAILED DESCRIPTION:
Primary objectives is: to compare exercise tolerance and aerobic capacity between healthy children with Bronchopulmonary Dysplasia children Only Bronchopulmonary Dysplasia children will realise the physical activity program.

Secondary objectives are: to analyse lung function and to evaluate flexibility.

ELIGIBILITY:
Bronchopulmonary Dysplasia Children

Inclusion Criteria:

* age between 4 to 6 years old
* Bronchopulmonary Dysplasia diagnostic
* ex-prematurity
* accept to participate.

Exclusion Criteria:

* congenital malformations
* neuromuscular disorders
* gait alterations
* difficulties for communication and understanding
* wheezing or pulmonary disease two weeks before to start the program
* hemodynamic changes (heart rate > 130bpm, systolic blood pressure > 130bpm, diastolic blood pressure > 80bpm).
* heart and/or lung transplantation.

Healthy children Criteria:

Inclusion Criteria:

* age between 4 to 6 years old.

Exclusion Criteria:

* antecedents of pulmonary or cardiac chronic disease
* congenital malformations
* neuromuscular disorders
* gait alterations
* difficulties for communication and understanding
* wheezing or pulmonary disease two weeks before to start the program
* hemodynamic changes (heart rate > 130bpm, systolic blood pressure > 130bpm, diastolic blood pressure > 80bpm).
* heart and/or lung transplantation.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
effort tolerance measured by six minute walking test | six minutes
aerobic capacity measured by shuttle run test | 15 minutes

SECONDARY OUTCOMES:
lung function measured by spirometry | 5 minutes
flexibility measured by sit and reach test | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Morales, Principal Investigator — Hospital de Nens de Barcelona
Locations (1):
- Hospital de Nens, Barcelona, Barcelona, Spain